CLINICAL TRIAL: NCT04147533
Title: A Prospective Phase II Clinical Trial Evaluating the Efficacy and the Safety of Tyrosine Kinase Inhibitors Withdrawal After a Previous Two-step Dose Reduction in Patients with Chronic Myeloid Leukemia in Deep Molecular Remission
Brief Title: Efficacy and Safety of TKIs' Withdrawal After a Two-step Dose Reduction in Patients with Chronic Myeloid Leukemia
Acronym: HALF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HALF2019
Record Dates: First submitted 2019-09-26; First posted 2019-11-01 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase; Withdrawal;Drug
Keywords: tyrosine kinase inhibitors; drug withdrawal; chronic myeloid leukemia, chronic phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Substance Withdrawal Syndrome | interventions — Dasatinib; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- initially treated patients (Experimental): The dose of tyrosin kinase inhibitors (imatinib, or nilotinib, or dasatinib) in patients meeting all of the inclusion criteria and none of the exclusion criteria will be reduced in two consequent steps, during the first 6 months after study entry by 50%, during the second 6 months by 50% again; the medication is discontinued then and the patients are followed each month in the first 6 months after withdrawal, each 1,5 month in the next 6 months, and each 3 months in the next 12 months.
  Interventions: Drug: Imatinib withdrawal; Drug: Dasatinib; Drug: Nilotinib

INTERVENTIONS:
Drug: Imatinib withdrawal — withdrawal of imatinib after previous two-step dose reduction: during the first 6 months after study entry, the dose of imatinib is 50% of the standard dose (200 mg daily), during the second 6 months after study entry, the dose of imatinib is 200 mg every other day; 12 months after study entry, imatinib is discontinued, the patient is followed in line with the aims of the trial
  Other Names: Glivec withdrawal
Drug: Dasatinib — withdrawal of dasatinib after previous two-step dose reduction: during the first 6 months after study entry, the dose of dasatinib is 50% of the standard dose (40 mg daily; tablets containing 50 mg are not available on the market), during the second 6 months after study entry, the dose of dasatinib is 40 mg every other day; 12 months after study entry, dasatinib is discontinued, the patient is followed in line with the aims of the trial
  Other Names: Sprycel withdrawal
Drug: Nilotinib — withdrawal of nilotinib after previous two-step dose reduction: during the first 6 months after study entry, the dose of nilotinib is 50% of the standard dose (200 mg every 12 hours), during the second 6 months after study entry, the dose of nilotinib is 400 mg every other day; 12 months after study entry, nilotinib is discontinued, the patient is followed in line with the aims of the trial
  Other Names: Tasigna withdrawal

SUMMARY:
Evaluation of the efficacy and safety of withdrawal of tyrosine kinase inhibitors after previous two-step dose reduction in patients with chronic myeloid leukemia in deep molecular remission

DETAILED DESCRIPTION:
In the first phase of the study (first 6 months after the study enrollment), 50% reduction of standard TKI dose follows.Physical and clinical examinations (focused on adverse effects and possible withdrawal syndrome manifestation) will be performed in predefined time intervals, pharmacological history of the subject will be taken, mandatory biochemical, hematological, and molecular-biological examinations will be performed.

In the following 6 months, the dose will be reduced by 50% i.e. medication will be administered every other day.

Twelve months after enrollment, the medication will be stoped. The subject is followed in predefined time intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented Ph1-positive and / or BCR-ABL1-positive CML in a documented first chronic phase, the criteria of which are as follows:

   * <15% blasts in peripheral blood (PB) or bone marrow (BM)
   * <30% blasts + promyelocytes in PB or BM
   * <20% of basophils in PB
   * >= 100 billion / l platelets
   * Absence of extramedullary involvement except hepato- and / or splenomegaly
2. Age >= 18 years
3. Signed informed consent to study participation
4. Typical [e13a2 (b2a2) or e14a2 (b3a2)] or atypical quantifiable type of BCR-ABL1 transcript on an international scale
5. Treatment of TKI either in the first line or in the second or other lines for intolerance only
6. TKI treatment> 4 years
7. Previous interferon-α treatment allowed with any treatment effect (intolerance / failure)
8. Deep molecular response >= MR4.0 lasting > 2 years
9. Participants in a fertile clinical trial must agree to use prescribed contraceptive methods from entry to study until one year after the last dose of study medication:

   * Women - Proper use of a highly reliable contraceptive method, ie combined hormonal contraceptives (in oral, vaginal or transdermal dosage form), gestagen hormonal contraceptives associated with ovulation inhibition (in oral or injectable dosage form), non-hormonal IUDs (intrauterine device) or IUDs , ev. presence of bilateral tubular occlusion, partner vasectomy, or adherence to sexual abstinence
   * Men - Observance of sexual abstinence or use of adequate contraceptive method (ie condom) in the case of sexual intercourse for the period from enrollment to 1 year after the last dose of the drug

Exclusion Criteria:

1. Patients with Ph1-positive and / or BCR-ABL1-positive CML in the second chronic phase, in the accelerated phase or blast crisis (AP/BC) at any time in the history of the disease
2. Non-quantifiable type of BCR-ABL1 transcript on an international scale
3. Treatment of TKI in the second or subsequent lines due to treatment failure according to ELN (European LeukemiaNet) criteria in 2006, 2009 or 2013
4. Previous failure of TKI treatment according to ELN criteria of 2006, 2009 or 2013
5. Previous allogeneic hematopoietic stem cell transplantation
6. Previous participation in a TKI withdrawal study with a real withdrawal history
7. Previous discontinuation of TKI outside the study for other reasons (eg intolerance or pregnancy) lasting more than 9 months and / or if a treatment response was lost during less than 12 months prior to screening
8. Life expectancy of less than 36 months due to severe concurrent disease
9. Severe concurrent disease that could limit adherence to study protocol or study completion
10. Pregnancy and breastfeeding
11. Disagreement or impossibility to comply with the contraceptive measures described in point 9 of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
proportion of patients in major molecular response, and MRFS at month 6 | 6 months after entry
  Proportion of patients in major molecular response (MMR) ie BCR-ABL1 (oncogenic BCR-ABL gene fusion) transcript levels <= 0.1%) and Molecular Recurrence-Free Survival (MRFS, ie time from study entry to MMR loss, ie BCR-ABL1 transcript levels > 0.1% in 2 consecutive samples, or death from any cause) at month 6 after study entry
proportion of patients in major molecular response (MMR) and MRFS at month 12 | 12 months after study entry
  Proportion of patients in major molecular response (MMR) and MRFS at month 12 after study entry
proportion of patients in MMR without treatment (TFR) and treatment-free survival at month 18 after study entry, ie. 6 months after treatment withdrawal | 18 months after study entry
  The proportion of patients in MMR without treatment (TFR) and treatment-free survival (TFS, ie the time from withdrawal of TKI (tyrosin kinase inhibitors) to loss of MMR, reinitiation of TKI therapy from any cause, progression, or death from any cause) at month 18 after study entry, ie, 6 months after treatment discontinuation
proportion of patients in MMR without treatment (TFR) and treatment-free survival at month 24 after study entry, ie. 12 months after treatment withdrawal | 24 months after study entry
  The proportion of patients in MMR without treatment (TFR) and treatment-free survival (TFS, ie the time from withdrawal of TKI to loss of MMR, reinitiation of TKI therapy from any cause, progression, or death from any cause) at month 24 after study entry, ie 12 months after treatment discontinuation
proportion of patients in MMR without treatment (TFR) and treatment-free survival at month 36 after study entry, ie. 24 months after treatment withdrawal | 36 months after study entry
  The proportion of patients in MMR without treatment (TFR) and treatment-free survival (TFS, ie the time from withdrawal of TKI to loss of MMR, reinitiation of TKI therapy from any cause, progression, or death from any cause) at month 36 after study entry, ie 24 months after treatment discontinuation

SECONDARY OUTCOMES:
Proportion of patients who lose MMR during de-escalation and in whom MMR and MR4.0 will recover after TKI re-introduction | every two months in the first 12 months, at early termination (due to pregnancy, investigator's,national competent authority's or sponsor's decision, poor adherence)
  Proportion of patients who lose MMR during de-escalation and in whom MMR and MR4.0 (deep molecular response, level of BCR-ABL transcripts <0.01% related to the international scale) will recover after TKI re-introduction
Proportion of patients who lose MMR after discontinuation of TKI and in whom MMR and MR4.0 will recover after TKI re-introduction | every month between month 13 and 18, every 1.5 month between month 18 and 24, every 3 months between month 24 and 36, at time of early termination
  Proportion of patients who lose MMR after discontinuation of TKI and in whom MMR and MR4.0 will recover after TKI re-introduction
Time to re-establish MMR and MR4.0 after TKI restart | since TKI restart until MMR and MR4.0 recovered (only in case that restart is necessary)
  Time to re-establish MMR and MR4.0 after TKI restart - evaluation every 3 months after TKI restart
Assessment of TKI's adverse effects dynamics during two-step reduction of their dose before withdrawal | every two months in the first 12 months, at early termination (due to pregnancy, investigator's,national competent authority's or sponsor's decision, poor adherence)
  Assessment of TKI's adverse effects dynamics during two-step reduction of their dose before withdrawal (using Common Terminology Criteria for Adverse Events; CTCAE classification with 5 grades)
Assessment of TKI withdrawal syndrome - proportion of patients with development of withdrawal syndrome | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Assessment of TKI withdrawal syndrome - proportion of patients with development of withdrawal syndrome) (using Common Terminology Criteria for Adverse Events; CTCAE classification with 5 grades)
Assessment of TKI withdrawal syndrome - severity of symptoms | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Assessment of TKI withdrawal syndrome - severity of symptoms (using Common Terminology Criteria for Adverse Events; CTCAE classification with 5 grades)
Assessment of TKI withdrawal syndrome - time to first complaint | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Assessment of TKI withdrawal syndrome - time to first complaint
Assessment of TKI withdrawal syndrome - duration of complaints | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Assessment of TKI withdrawal syndrome - duration of complaints
Assessment of TKI withdrawal syndrome - therapeutic intervention | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Assessment of TKI withdrawal syndrome - therapeutic intervention (pharmacological history, dose changes)
Assessment of the correlation between adverse effects on previous TKI treatment and possible withdrawal syndrome | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Assessment of the correlation between adverse effects on previous TKI treatment and possible withdrawal syndrome (using Common Terminology Criteria for Adverse Events; CTCAE classification with 5 grades)
BCR-ABL1 kinetics during TKI therapy | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  number of BCR-ABL1 transcripts during TKI therapy
Correlation of BCR-ABL1 kinetics (number of BCR-ABL1 transcripts in time) during TKI therapy with potential molecular relapse after TKI discontinuation | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Correlation of BCR-ABL1 kinetics during TKI therapy with potential molecular relapse after TKI discontinuation
Correlation of the effect of TKI dose reduction and subsequent discontinuation with lipid metabolism and glycemia (using Common Terminology Criteria for Adverse Events; CTCAE classification with 5 grades) | months 2,4,6,8,10,12,15,18,21,24,30,36
  Correlation of the effect of TKI dose reduction and subsequent discontinuation with lipid metabolism and glycemia (using Common Terminology Criteria for Adverse Events; CTCAE classification with 5 grades)

OTHER OUTCOMES:
failure-free survival | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  failure-free survival
progression-free survival | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  progression-free survival
overall survival | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  overall survival
Assessment of correlation of age with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of age with success of TFR / survival without molecular recurrence
Assessment of correlation of gender with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of gender with success of TFR / survival without molecular recurrence
Assessment of correlation of Sokal index (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of Sokal index (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence
Assessment of correlation of Hasford score (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of Hasford score (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence
Assessment of correlation of EUTOS score (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of EUTOS score (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence
Assessment of correlation of ELTS score (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of ELTS score (calculated in time of diagnosis; if available) with success of TFR / survival without molecular recurrence
Assessment of correlation of BCR-ABL1 transcript type with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of BCR-ABL1 transcript type with success of TFR / survival without molecular recurrence
Assessment of correlation of previous interferon alfa therapy (yes/no) with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of previous interferon alfa therapy (yes/no) with success of TFR / survival without molecular recurrence
Assessment of correlation of previous interferon alfa therapy length with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of previous interferon alfa therapy length with success of TFR / survival without molecular recurrence
Assessment of correlation of TKI type - imatinib - with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of TKI type - imatinib - with success of TFR / survival without molecular recurrence
Assessment of correlation of TKI type - nilotinib - with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of TKI type - nilotinib - with success of TFR / survival without molecular recurrence
Assessment of correlation of TKI type - dasatinib - with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of TKI type - dasatinib - with success of TFR / survival without molecular recurrence
Assessment of correlation of length of imatinib therapy prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of length of imatinib therapy prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of length of dasatinib therapy prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of length of dasatinib therapy prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of length of nilotinib therapy prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of length of nilotinib therapy prior to study entry with success of TFR / survival without molecular recurrence
Plasma concentration of imatinib prior to study entry | day 0
  Plasma concentration of imatinib prior to study entry
Plasma concentration of imatinib during dose deescalation period | month 6, 12
  Plasma concentration of imatinib during dose deescalation period
Plasma concentration of nilotinib prior to study entry | day 0
  Plasma concentration of nilotinib prior to study entry
Plasma concentration of nilotinib during dose deescalation period | month 6, 12
  Plasma concentration of nilotinib during dose deescalation period
Plasma concentration of dasatinib prior to study entry | day 0
  Plasma concentration of dasatinib prior to study entry
Plasma concentration of dasatinib during dose deescalation period | month 6, 12
  Plasma concentration of dasatinib during dose deescalation period
Assessment of correlation of imatinib plasma concentration during dose deescalation period with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of imatinib plasma concentration during dose deescalation period with success of TFR / survival without molecular recurrence
Assessment of correlation of imatinib plasma concentration prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of imatinib plasma concentration prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of nilotinib plasma concentration prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of nilotinib plasma concentration prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of nilotinib plasma concentration during dose deescalation period with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of nilotinib plasma concentration during dose deescalation period with success of TFR / survival without molecular recurrence
Assessment of correlation of dasatinib plasma concentration prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of dasatinib plasma concentration prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of dasatinib plasma concentration during dose deescalation period with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of dasatinib plasma concentration during dose deescalation period with success of TFR / survival without molecular recurrence
Assessment of correlation of time needed to establish DMR after TKI start with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of time needed to establish DMR after TKI start with success of TFR / survival without molecular recurrence
Assessment of correlation of deep molecular response length prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of deep molecular response length prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of molecular response depth (MMR i.e. BCR-ABL1<=0,1% vs. DMR i.e. BCR-ABL1<=0,01%) at study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of molecular response depth (major molecular response i.e. BCR-ABL1<=0,1% vs. deep molecular response i.e. BCR-ABL1<=0,01%) at study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of molecular response depth (major molecular response i.e. BCR-ABL1<=0,1% vs. deep molecular response i.e. BCR-ABL1<=0,01%) at TKI discontinuation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of molecular response depth (major molecular response i.e. BCR-ABL1<=0,1% vs. deep molecular response i.e. BCR-ABL1<=0,01%) at TKI discontinuation with success of TFR / survival without molecular recurrence
Assessment of correlation of early molecular response (BCR-ABL1 transcript levels at month 3 of TKI treatment ≤ 10% versus > 10%) with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of early molecular response (BCR-ABL1 transcript levels at month 3 of TKI treatment ≤ 10% versus > 10%) with success of TFR / survival without molecular recurrence
Assessment of correlation of withdrawal syndrome with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of withdrawal syndrome (using CTCAE 5 grade classification) with success of TFR / survival without molecular recurrence
Assessment of correlation of white blood cells number in leukocyte subpopulations in peripheral blood prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of white blood cells number in leukocyte subpopulations in peripheral blood prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of white blood cells activation in leukocyte subpopulations in peripheral blood(defined below The immunological profile of patients with CML) prior to study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of white blood cells activation in leukocyte subpopulations in peripheral blood(defined below The immunological profile of patients with CML) prior to study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of white blood cells number in leukocyte subpopulations in peripheral blood during TKI dose deescalation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of white blood cells number in leukocyte subpopulations in peripheral blood during TKI dose deescalation with success of TFR / survival without molecular recurrence
Assessment of correlation of white blood cells activation in leukocyte subpopulations in peripheral blood during TKI dose deescalation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of white blood cells activation in leukocyte subpopulations in peripheral blood (defined below The immunological profile of patients with CML) during TKI dose deescalation with success of TFR / survival without molecular recurrence
Assessment of correlation of white blood cells number in leukocyte subpopulations in peripheral blood after TKI discontinuation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of white blood cells number in leukocyte subpopulations in peripheral blood during TKI dose deescalation with success of TFR / survival without molecular recurrence
Assessment of correlation of white blood cells activation in leukocyte subpopulations in peripheral blood after TKI discontinuation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of white blood cells activation in leukocyte subpopulations in peripheral blood (defined below The immunological profile of patients with CML) after TKI discontinuation with success of TFR / survival without molecular recurrence
Assessment of correlation of minimal residual disease at the DNA level (gBCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) at study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of minimal residual disease at the DNA level (gBCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) at study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of minimal residual disease at the DNA level (gBCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) during TKI dose deescalation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of minimal residual disease at the DNA level (gBCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) during TKI dose deescalation with success of TFR / survival without molecular recurrence
Assessment of correlation of minimal residual disease at the DNA level (gBCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) after TKI discontinuation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of minimal residual disease at the DNA level (gBCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) after TKI discontinuation with success of TFR / survival without molecular recurrence
Assessment of correlation of minimal residual disease at the mRNA level (BCR-ABL1) using digital PCR (ddPCR) at study entry with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of minimal residual disease at the mRNA level (BCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) at study entry with success of TFR / survival without molecular recurrence
Assessment of correlation of minimal residual disease at the mRNA level (BCR-ABL1) using digital PCR (ddPCR) during TKI dose deescalation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of minimal residual disease at the mRNA level (BCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) during TKI dose deescalation with success of TFR / survival without molecular recurrence
Assessment of correlation of minimal residual disease at the mRNA level (BCR-ABL1) using digital PCR (ddPCR) after TKI discontinuation with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of minimal residual disease at the mRNA level (BCR-ABL1) using digital PCR (ddPCR) (see below Quantification of minimal residual disease) after TKI discontinuation with success of TFR / survival without molecular recurrence
Assessment of correlation of gene promoters' genotypes coding transmembrane imatinib transporters with success of TFR / survival without molecular recurrence | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of gene promoters' genotypes coding transmembrane imatinib transporters (genes SLC22A4, SLC22A5) (see below Genotype analysis of imatinib transmembrane transporter gene promoters) with success of TFR / survival without molecular recurrence
The immunological profile of patients with CML (characteristics of lymphocyte subpopulations in peripheral blood - cells number) prior to study entry | baseline
  The immunological profile of patients with CML (analysis of lymphocyte subpopulations - number of T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood) prior to study entry
Correlation of characteristics of lymphocyte subpopulations in peripheral blood - cells number in peripheral blood with frequency of the withdrawal syndrome prior to study entry | baseline
  Correlation of characteristics of lymphocyte subpopulations in peripheral blood - T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood with frequency of the withdrawal syndrome prior to study entry
Correlation of characteristics of lymphocyte subpopulations in peripheral blood - cells number in peripheral blood with severity of the withdrawal syndrome prior to study entry | baseline
  Correlation of characteristics of lymphocyte subpopulations in peripheral blood - T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood with severity of the withdrawal syndrome prior to study entry
The immunological profile of patients with CML (characteristics of lymphocyte subpopulations in peripheral blood - cells number) during TKI dose deescalation | month 6,12
  The immunological profile of patients with CML (analysis of lymphocyte subpopulations - number of T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood) during TKI dose deescalation
Correlation of characteristics of lymphocyte subpopulations in peripheral blood - cells number in peripheral blood with frequency of the withdrawal syndrome during TKI dose deescalation | month 6,12
  Correlation of characteristics of lymphocyte subpopulations in peripheral blood - T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood with frequency of the withdrawal syndrome during TKI dose deescalation
Correlation of characteristics of lymphocyte subpopulations in peripheral blood - cells number in peripheral blood with severity of the withdrawal syndrome during TKI dose deescalation | month 6,12
  Correlation of characteristics of lymphocyte subpopulations in peripheral blood - T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood with severity of the withdrawal syndrome during TKI dose deescalation
The immunological profile of patients with CML (characteristics of lymphocyte subpopulations in peripheral blood - cells number) after TKI discontinuation | month 24
  The immunological profile of patients with CML (analysis of lymphocyte subpopulations - number of T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood) after TKI discontinuation
Correlation of characteristics of lymphocyte subpopulations in peripheral blood - cells number in peripheral blood with frequency of the withdrawal syndrome after TKI discontinuation | month 24
  Correlation of characteristics of lymphocyte subpopulations in peripheral blood - T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood with frequency of the withdrawal syndrome after TKI discontinuation
Correlation of characteristics of lymphocyte subpopulations in peripheral blood - cells number in peripheral blood with the severity of the withdrawal syndrome after TKI discontinuation | month 24
  Correlation of characteristics of lymphocyte subpopulations in peripheral blood - T-lymphocytes (T-ly), CD4-T-lymphocytes, CD8T-lymphocytes, T-regulatory-lymphocytes (CD 3+4+25+127-), B-lymphocytes, Natural-Killer-Cells number, myeloid-derived suppressor cells in peripheral blood with severity of the withdrawal syndrome after TKI discontinuation
Quantification of minimal residual disease using the highly sensitive ddPCR method at the DNA level using patient-specific BCR-ABL1 gene fusions | day 0, months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Quantification of minimal residual disease using the highly sensitive ddPCR (digital polymerase chain reaction) method at the DNA level using patient-specific BCR-ABL1 gene fusions
Creating a mathematic predictive model to predict TFR by the minimal residual disease (defined by the highly sensitive ddPCR method at the DNA level using patient-specific BCR-ABL1 gene fusions) | day 0, months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Creating a mathematic predictive model to predict TFR by the minimal residual disease (defined by the highly sensitive ddPCR method at the DNA level using patient-specific BCR-ABL1 gene fusions)
Quantification of minimal residual disease using the highly sensitive ddPCR method at BCR-ABL1 mRNA level | day 0, months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Quantification of minimal residual disease using the highly sensitive ddPCR method at BCR-ABL1 mRNA (messenger RNA) level
Creating a mathematic predictive model to predict TFR by the minimal residual disease (defined by the highly sensitive ddPCR method at BCR-ABL1 mRNA level) | day 0, months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Creating a mathematic predictive model to predict TFR by the minimal residual disease (defined by the highly sensitive ddPCR method at BCR-ABL1 mRNA level)
Genotype analysis of imatinib transmembrane transporter gene promoters SLC22A4 | baseline
  Genotype analysis of imatinib transmembrane transporter gene promoters SLC22A4 (Solute carrier family 22, member 4)
Genotype analysis of imatinib transmembrane transporter gene promoters SLC22A5 | baseline
  Genotype analysis of imatinib transmembrane transporter gene promoters SLC22A5 (Solute carrier family 22 member 5)
Creating a mathematical predictive model to predict a molecular relapse using BCR-ABL1 transcripts levels kinetics during TKI administration (see above BCR-ABL1 kinetics during TKI therapy) | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Creating a mathematical predictive model to predict a molecular relapse using BCR-ABL1 transcripts levels kinetics during TKI administration (see above BCR-ABL1 kinetics during TKI therapy)
Analysis of molecular mutations within clonal hematopoiesis using NGS | baseline
  Analysis of molecular mutations within clonal hematopoiesis using NGS (new generation sequencing) - panel of mutations of interest: ASXL1, RUNX1, TET2, DNMT3A, NRAS, TP53, JAK2, BCOR, EZH2, CBL, ZRSR2, IDH1, U2AF (PTPN11, U2AF1
Assessment of correlation of molecular mutations occurrence within clonal hematopoiesis (using NGS) with TFR / molecular recurrence-free survival | months 2,4,6,8,10,12,15,18,21,24,30,36
  Assessment of correlation of molecular mutations occurrence within clonal hematopoiesis (using NGS) with TFR / molecular recurrence-free survival
Evaluation of economic aspects of TKI dose reduction (cost benefit analysis) | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Evaluation of economic aspects of TKI dose reduction (cost benefit analysis)
Evaluation of economic aspects of TKI discontinuation (cost benefit analysis) | months 2,4,6,8,10,12,13,14,15,16,17,18,19.5,21,22.5,24,27,30,33,36
  Evaluation of economic aspects of TKI discontinuation (cost benefit analysis)
Assessing the proportion of patients entering the study out of the total number of patients meeting the study entry criteria | day -28-0
  Assessing the proportion of patients entering the study out of the total number of patients meeting the study entry criteria
Quality of life assessment during dose de-escalation and after TKI discontinuation - Do you have any trouble doing strenuous activities, like carrying a heavy shopping bag or a suitcase? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Do you have any trouble doing strenuous activities, like carrying a heavy shopping bag or a suitcase? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Do you have any trouble taking a long walk? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Do you have any trouble taking a long walk? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Do you have any trouble taking a short walk outside of the house? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Do you have any trouble taking a short walk outside of the house? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Do you need to stay in bed or a chair during the day? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Do you need to stay in bed or a chair during the day? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Do you need help with eating, dressing, washing yourself or using the toilet? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Do you need help with eating, dressing, washing yourself or using the toilet? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Were you limited in doing either your work or other daily activities? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Were you limited in doing either your work or other daily activities? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Were you limited in pursuing your hobbies or other leisure time activities? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Were you limited in pursuing your hobbies or other leisure time activities? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Were you short of breath? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Were you short of breath? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had pain? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you had pain? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Did you need to rest? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Did you need to rest? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had trouble sleeping? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you had trouble sleeping? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you felt weak? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you felt weak? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you lacked appetite? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you lacked appetite? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you felt nauseated? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you felt nauseated? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you vomited? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you vomited? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you been constipated? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you been constipated? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had diarrhea? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you had diarrhea? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Were you tired? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Were you tired? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Did pain interfere with your daily activities? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Did pain interfere with your daily activities? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had difficulty in concentrating on things, like reading a newspaper or watching television? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you had difficulty in concentrating on things, like reading a newspaper or watching television? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Did you feel tense? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Did you feel tense? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Did you worry? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Did you worry? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Did you feel irritable? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Did you feel irritable? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Did you feel depressed? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Did you feel depressed? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had difficulty remembering things? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Have you had difficulty remembering things? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Has your physical condition or medical treatment interfered with your family life? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Has your physical condition or medical treatment interfered with your family life? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Has your physical condition or medical treatment interfered with your social activities? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Has your physical condition or medical treatment interfered with your social activities? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Has your physical condition or medical treatment caused you financial difficulties? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - Has your physical condition or medical treatment caused you financial difficulties? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - How would you rate your overall health during the past week? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - How would you rate your overall health during the past week? 1 (very poor) -2-3-4-5-6-7 (excellent)
Quality of life assessment during dose de-escalation and after TKI discontinuation - How would you rate your overall quality of life during the past week? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-C30) - How would you rate your overall quality of life during the past week? 1 (very poor) -2-3-4-5-6-7 (excellent)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had abdominal pains or cramps? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had abdominal pains or cramps? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had a dry mouth? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had a dry mouth? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you been concerned about changes in your weight? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you been concerned about changes in your weight? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had skin problems (e.g. color changes, itchy, dry or flaking skin)? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had skin problems (e.g. color changes, itchy, dry or flaking skin)? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had headaches? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had headaches? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had aches or pains in your muscles or joints? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had aches or pains in your muscles or joints? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had hair loss? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had hair loss? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you sweated? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you sweated? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had acid indigestion or heartburn? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had acid indigestion or heartburn? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you felt drowsy? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you felt drowsy? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you experienced any swelling in certain parts of your body (e.g. ankles, legs or around your eyes)? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you experienced any swelling in certain parts of your body (e.g. ankles, legs or around your eyes)? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had to urinate frequently? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had to urinate frequently? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had problems with your eyes (e.g. burning, watery, irritated or dry)? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had problems with your eyes (e.g. burning, watery, irritated or dry)? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had muscle cramps? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had muscle cramps? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had emotional ups and downs? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had emotional ups and downs? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you worried about your future health? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you worried about your future health? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you had any difficulties carrying on with your usual activities because of getting tired easily? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you had any difficulties carrying on with your usual activities because of getting tired easily? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you worried about getting an infection? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you worried about getting an infection? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you felt dissatisfied with your body as result of the disease or treatment? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you felt dissatisfied with your body as result of the disease or treatment? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - How much has your treatment been a burden to you? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - How much has your treatment been a burden to you? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you needed social support (e.g. family, friends or relatives) to undergo therapy or to cope with the disease? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you needed social support (e.g. family, friends or relatives) to undergo therapy or to cope with the disease? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you felt satisfied with the care you have received? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you felt satisfied with the care you have received? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you felt satisfied with the information you have received (e.g. about the disease and its treatment)? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you felt satisfied with the information you have received (e.g. about the disease and its treatment)? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)
Quality of life assessment during dose de-escalation and after TKI discontinuation - Have you felt satisfied with the quality of your social life (including family and/ or friends)? | day 0, month 6,12,18, 24, 36
  Quality of life assessment during dose de-escalation and after TKI discontinuation (using EORTC questionnaires QLQ-CML24) - Have you felt satisfied with the quality of your social life (including family and/ or friends)? not at all (1 point) - a little (2 points) - quite a bit (3 points) - very much (4 points)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Zackova, Principal Investigator — University Hospital Brno
Locations (8):
- Czechia (8):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - University Hospital Plzen, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
  - Insitute of Hematology and Blood Transfusion, Prague
  - General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: No